CLINICAL TRIAL: NCT00000177
Title: Estrogen Hormone Protocol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: IA0001; 3U01AG010483-08S2 (NIH)
Record Dates: First submitted 1999-10-29; First posted 1999-11-01 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-09

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; Estrogen
MeSH Terms: conditions — Alzheimer Disease | interventions — Estrogens

INTERVENTIONS:
Drug: Estrogen

SUMMARY:
Estrogen is a hormone that is dominant in the female reproductive system. In women, most estrogen is produced by the ovaries. Men produce estrogen by converting testosterone into estrogen. Because this hormone also has many beneficial effects on brain cells, it currently is being studied as a treatment for Alzheimer's disease. The enzyme that forms the neurotransmitter acetylcholine is promoted in the presence of estrogen. Several very small clinical studies have demonstrated improvement in cognitive function and mood measures in women with Alzheimer's disease who take estrogen.

ELIGIBILITY:
Inclusion Criteria:

* Women with a diagnosis of Alzheimer's disease who currently are not taking estrogen replacement therapy, who have had a hysterectomy, and who are in stable general health.

Exclusion Criteria:

* Patients with an uncontrolled health problem, such as untreated high blood pressure or thyroid disease.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 1995-10; Primary Completion 1999-01 (Actual); Study Completion 1999-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon Thal, MD., Principal Investigator — University of California, San Diego
Locations (25):
- United States (25):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California, San Diego, San Diego, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Rush Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - New York University Medical Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - Burke Medical Research Institute, White Plains, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Result] Mulnard RA, Cotman CW, Kawas C, van Dyck CH, Sano M, Doody R, Koss E, Pfeiffer E, Jin S, Gamst A, Grundman M, Thomas R, Thal LJ. Estrogen replacement therapy for treatment of mild to moderate Alzheimer disease: a randomized controlled trial. Alzheimer's Disease Cooperative Study. JAMA. 2000 Feb 23;283(8):1007-15. doi: 10.1001/jama.283.8.1007. PMID 10697060
- See also: The Alzheimer's Disease Education and Referral (ADEAR) Center is a service of the National Institute on Aging (NIA). — http://www.adcs.org/